CLINICAL TRIAL: NCT05200156
Title: The Impact Of Choline Administration On Oxidative Stress And Clinical Outcome Of Patients With Non-Alcoholic Fatty Liver Disease NAFLD
Brief Title: Impact Of Choline in Patients With NAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amal A. Elkholy, Lecturer of Clinical Pharmacy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Choline in NAFLD
Record Dates: First submitted 2021-11-17; First posted 2022-01-20 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Choline and Leptin/Thiobarbituric acid reactive substances
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Phosphatidylcholines

STUDY DESIGN:
Intervention Model Description: The study is a Prospective, Randomized, Controlled, single blinded study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Choline supplement group (Experimental): Phosphatidyl choline tablets at a dose of 1200 mg twice per day plus conventional management for 12 weeks
  Interventions: Dietary Supplement: Phosphatidyl Choline
- Control group (No Intervention): conventional management only for 12 weeks

INTERVENTIONS:
Dietary Supplement: Phosphatidyl Choline — conventional management + phosphatidyl choline tablets
  Arms: Choline supplement group

SUMMARY:
The study will be assessing the impact of choline supplementation in Non-alcoholic fatty liver disease patients using ultrasonography to show change in liver echogenicity, various laboratory tests as liver function, lipid profile and glucose control tests and finally on markers of oxidative stress as Thiobarbituric acid reactive substances and Leptin.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) has attracted increasing attention given its high prevalence, estimated at 20% to 44% in Western countries and 5% to 38% in Asia as well as its correlation with cardiovascular morbidity and mortality.

NAFLD is the result of hepatic fat accumulation in patients without a history of excessive alcohol consumption, predisposing medications or other defined liver disorders. NAFLD comprises a spectrum of liver disorders. At one end of this spectrum, is simple hepatic steatosis and the other end is non-alcoholic steatohepatitis (NASH) which is characterized by hepatocellular injury, inflammation and fibrosis sometimes leading to cirrhosis. It is considered the hepatic manifestation of metabolic syndrome, which is defined by the presence of central obesity, insulin resistance, hyperlipidemia, hyperglycemia, and hypertension.

According to the multiple parallel hits in NAFLD pathogenesis, the first hit is insulin resistance, which results in increased hepatic de novo lipogenesis and impaired adipose tissue lipolysis.These conditions cause an efflux of free fatty acids from the adipose tissue to the liver. The liver becomes vulnerable to a series of hits, including oxidative stress and dysregulation of adipokines such as leptin.

It has been also observed that fatty liver can occur both in people with a normal body mass index (BMI) (10-24% of the population has fatty liver) and in 95% of adults with obesity.

Choline is an essential nutrient for human health, which exerts various physiological functions:

1. It is acetylated to generate acetylcholine, the important neurotransmitter;
2. It is oxidized to pass methyl to S-adenosylmethionine, a universal methyl group donor, which participates in the methylation-dependent biosynthesis of DNA, RNA and protein;
3. It is phosphorylated to synthesize phosphatidylcholine, a major constituent of cell and mitochondrial membranes, which is involved in the mitochondrial bioenergetics regulating lipid and glucose metabolism. In addition, it takes part in the packaging and exporting of triglyceride (TG) in very low-density lipoprotein (VLDL), as well as the solubilizing of bile salts for secretion.

Choline deficiency contributes to various disorders in animals and humans, with liver as its main target. Humans deprived of choline have been perceived to develop fatty liver, liver cell death or skeletal muscle damage, which were further proven by another clinical study revealing that patients fed with total parenteral nutrition (TPN) solutions low in choline resulted in TPN-associated liver disease.

Growing evidence has suggested certain effects of choline on mitochondrial metabolism. Low choline results in the altered composition of mitochondrial membranes, reduced mitochondrial membrane potential, decreased Adenosine triphosphate production and disturbance in fatty acid β-oxidation in rats fed a choline-deficient diet. This mitochondrial dysfunction has also been linked to the process of the increase of reactive oxygen species (ROS) generation, the loss of mitochondrial membrane potential, cellular apoptosis and hepatocarcinogenesis caused by choline deficiency in rat hepatocytes. However, the specific mechanisms connecting choline, DNA methylation and metabolic diseases, such as non-alcoholic fatty liver disease (NAFLD), remain to be evidently described.

Excessive energy substrates available to the hepatocytes can potentially result in cellular steatosis with the increasing generation of free fatty acids (FFA) and ROS, which, in turn, will lead to mitochondrial dysfunction inseparably linked with oxidative stress. This is fundamental to the development of dietary-induced NAFLD or TPN-associated liver disease under unbalanced nutrients distress and can potentially lead to steatohepatitis, fibrosis and cirrhosis in the liver.

Considering those mechanisms, hence it is interesting to study whether supplementation of choline could have a potential benefit in NAFLD patients. Choline has been shown to decrease lipoprotein oxidation, generation of inflammatory mediators and reactive oxygen species, maintain lipid and glucose homeostasis and help in the repair of mitochondrial membrane.

Patients with NAFLD exhibit increased levels of hepatic cytochrome P450-2E1 and thiobarbituric acid reactants, which are markers of lipid peroxidation. Oxidative stress has been demonstrated in animal and human studies to be a significant factor, responsible for causing progression of NAFLD to NASH. In this respect, it may be regarded as an important second hit.

Oxidative stress in fatty liver arises because of excessive fatty acid oxidation resulting in an increase release of reactive oxygen species. Another study demonstrated that, total lipid peroxidation products as represented by TBARS were significantly higher among patients with NAFLD as compared to patients with either chronic viral hepatitis or healthy controls.

This suggests that the occurrence of high plasma concentration of products of lipid peroxidation is a unique phenomenon in patients with NAFLD and not only a byproduct of any inflammation, because TBARS was lower among patients with chronic viral hepatitis who had high degree of necroinflammation.

Leptin, an important regulatory energy hormone, is released from adipocytes and may play a role in the development of liver steatosis. High levels of serum leptin have been reported in patients with NAFLD.

Although the underlying mechanisms of leptin in NAFLD are incompletely understood, it has been suggested that it affects fat deposition, fibrogenesis, and inflammation in the liver of patients with NAFLD.

In NAFLD, the dysregulation of adipokines, including leptin, mediate insulin resistance through reduced insulin signaling, increased fatty acid concentrations in the liver, and promote steatosis.In addition to hyperinsulinemia, a feature of insulin resistance is the stimulatory effect on the leptin gene, which causes the release of leptin in a vicious cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Patients from 18 to 65 years.
2. Gender: both males and females (age and sex matched in both groups).
3. Patients diagnosed with NAFLD via ultrasound (hepatic steatosis observation on ultrasound).
4. Treatment free from choline supplementation for the past 3 months prior starting the therapeutic regimen.

Exclusion Criteria:

1. Other liver diseases as viral hepatitis (B or C)
2. Alcohol consumption more than 40 g per week for the past 12 months, and life-time cumulative consumption more than 100 kg.
3. Autoimmune liver disease
4. Malignancy of any nature.
5. Any systemic failure (cardiovascular, renal or respiratory)
6. Patients with major psychiatric illness.
7. Pregnant or lactating women.
8. Diabetes mellitus .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
effect on Oxidative stress marker as the mean change of Thiobarbituric acid reactive substances level | 12 weeks
  Measured as the mean change in Thiobarbituric acid reactive substances serum level (mmol/μg) at baseline and after 12 weeks of choline supplementation

SECONDARY OUTCOMES:
effect on Inflammatory status as the mean change in leptin levels | 12 weeks
  Measured by Inflammation marker as the mean change in serum leptin levels (ng/mL) at baseline and after 12 weeks of choline supplementation

OTHER OUTCOMES:
Clinical outcome as measured by Hepatic ultrasonography | 12 weeks
  ultrasonography measure the change in liver size at baseline and after 12 weeks.
Clinical outcome as measured by Hepatic US | 12 weeks
  ultrasonography measure the change in echogenicity at baseline and after 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Lamia El Wakeel, PhD, Principal Investigator — Ain Shams University; Doaa Zakaria, PhD, Principal Investigator — Ain Shams University
Locations (1):
- Tropical Medicine Department, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lockman KA, Baren JP, Pemberton CJ, Baghdadi H, Burgess KE, Plevris-Papaioannou N, Lee P, Howie F, Beckett G, Pryde A, Jaap AJ, Hayes PC, Filippi C, Plevris JN. Oxidative stress rather than triglyceride accumulation is a determinant of mitochondrial dysfunction in in vitro models of hepatic cellular steatosis. Liver Int. 2012 Aug;32(7):1079-92. doi: 10.1111/j.1478-3231.2012.02775.x. Epub 2012 Mar 19. PMID 22429485
- [Background] Bahrami M, Cheraghpour M, Jafarirad S, Alavinejad P, Asadi F, Hekmatdoost A, Mohammadi M, Yari Z. The effect of melatonin on treatment of patients with non-alcoholic fatty liver disease: a randomized double blind clinical trial. Complement Ther Med. 2020 Aug;52:102452. doi: 10.1016/j.ctim.2020.102452. Epub 2020 May 23. PMID 32951715
- [Background] Buchman AL. The addition of choline to parenteral nutrition. Gastroenterology. 2009 Nov;137(5 Suppl):S119-28. doi: 10.1053/j.gastro.2009.08.010. PMID 19874943
- [Background] Canbakan B, Tahan V, Balci H, Hatemi I, Erer B, Ozbay G, Sut N, Hacibekiroglu M, Imeryuz N, Senturk H. Leptin in nonalcoholic fatty liver disease. Ann Hepatol. 2008 Jul-Sep;7(3):249-54. PMID 18753993
- [Background] Corbin KD, Zeisel SH. Choline metabolism provides novel insights into nonalcoholic fatty liver disease and its progression. Curr Opin Gastroenterol. 2012 Mar;28(2):159-65. doi: 10.1097/MOG.0b013e32834e7b4b. PMID 22134222
- [Background] Guo WX, Pye QN, Williamson KS, Stewart CA, Hensley KL, Kotake Y, Floyd RA, Broyles RH. Mitochondrial dysfunction in choline deficiency-induced apoptosis in cultured rat hepatocytes. Free Radic Biol Med. 2005 Sep 1;39(5):641-50. doi: 10.1016/j.freeradbiomed.2005.04.013. PMID 16085182
- [Background] Hassan K, Bhalla V, El Regal ME, A-Kader HH. Nonalcoholic fatty liver disease: a comprehensive review of a growing epidemic. World J Gastroenterol. 2014 Sep 14;20(34):12082-101. doi: 10.3748/wjg.v20.i34.12082. PMID 25232245
- [Background] Lee JH, Kim D, Kim HJ, Lee CH, Yang JI, Kim W, Kim YJ, Yoon JH, Cho SH, Sung MW, Lee HS. Hepatic steatosis index: a simple screening tool reflecting nonalcoholic fatty liver disease. Dig Liver Dis. 2010 Jul;42(7):503-8. doi: 10.1016/j.dld.2009.08.002. Epub 2009 Sep 18. PMID 19766548
- [Background] Madan K, Bhardwaj P, Thareja S, Gupta SD, Saraya A. Oxidant stress and antioxidant status among patients with nonalcoholic fatty liver disease (NAFLD). J Clin Gastroenterol. 2006 Nov-Dec;40(10):930-5. doi: 10.1097/01.mcg.0000212608.59090.08. PMID 17063114
- [Background] Mishra A, Younossi ZM. Epidemiology and Natural History of Non-alcoholic Fatty Liver Disease. J Clin Exp Hepatol. 2012 Jun;2(2):135-44. doi: 10.1016/S0973-6883(12)60102-9. Epub 2012 Jul 21. PMID 25755422
- [Background] Mirza MS. Obesity, Visceral Fat, and NAFLD: Querying the Role of Adipokines in the Progression of Nonalcoholic Fatty Liver Disease. ISRN Gastroenterol. 2011;2011:592404. doi: 10.5402/2011/592404. Epub 2011 Aug 28. PMID 21991518
- [Background] Polyzos SA, Kountouras J, Mantzoros CS. Leptin in nonalcoholic fatty liver disease: a narrative review. Metabolism. 2015 Jan;64(1):60-78. doi: 10.1016/j.metabol.2014.10.012. Epub 2014 Oct 23. PMID 25456097
- [Background] Sanyal AJ, Campbell-Sargent C, Mirshahi F, Rizzo WB, Contos MJ, Sterling RK, Luketic VA, Shiffman ML, Clore JN. Nonalcoholic steatohepatitis: association of insulin resistance and mitochondrial abnormalities. Gastroenterology. 2001 Apr;120(5):1183-92. doi: 10.1053/gast.2001.23256. PMID 11266382
- [Background] Yesilova Z, Yaman H, Oktenli C, Ozcan A, Uygun A, Cakir E, Sanisoglu SY, Erdil A, Ates Y, Aslan M, Musabak U, Erbil MK, Karaeren N, Dagalp K. Systemic markers of lipid peroxidation and antioxidants in patients with nonalcoholic Fatty liver disease. Am J Gastroenterol. 2005 Apr;100(4):850-5. doi: 10.1111/j.1572-0241.2005.41500.x. PMID 15784031
- [Background] Younossi Z, Anstee QM, Marietti M, Hardy T, Henry L, Eslam M, George J, Bugianesi E. Global burden of NAFLD and NASH: trends, predictions, risk factors and prevention. Nat Rev Gastroenterol Hepatol. 2018 Jan;15(1):11-20. doi: 10.1038/nrgastro.2017.109. Epub 2017 Sep 20. PMID 28930295
- [Background] Zeisel SH. Choline: critical role during fetal development and dietary requirements in adults. Annu Rev Nutr. 2006;26:229-50. doi: 10.1146/annurev.nutr.26.061505.111156. PMID 16848706
- [Derived] Sedhom SS, El Wakeel LM, Barakat EMF, Shousha HI, Shamkh MA, Salama SH, Zaky DZ, El Kholy AA. The impact of choline supplementation on oxidative stress and clinical outcomes among patients with non-alcoholic fatty liver disease: a randomized controlled study. Ther Adv Chronic Dis. 2025 Aug 17;16:20406223251358659. doi: 10.1177/20406223251358659. eCollection 2025. PMID 40838115